CLINICAL TRIAL: NCT06587984
Title: Influenza Reminder Text-Messaging: A Randomized Quality Improvement Effort to Promote Influenza Vaccine in Pediatric Primary Care
Brief Title: Influenza Reminder Text-Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 24-022516
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients (recipients of text message reminders) will not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1a (No Intervention): Patients within Cohort 1 have an upcoming well child visit between September-December 2024. Patients within Cohort 1a are those randomized to CONTROL and will not receive a text message reminder about getting their flu shot at their upcoming visit.
- Cohort 1b (Experimental): Patients within Cohort 1 have an upcoming well child visit between September-December 2024. Patients within Cohort 1b are those randomized to INTERVENTION MESSAGE #1 and will receive text message reminder (variation #1) about getting their flu shot at their upcoming visit.
  Interventions: Behavioral: Text message reminder
- Cohort 1c (Experimental): Patients within Cohort 1 have an upcoming well child visit between September-December 2024. Patients within Cohort 1c are those randomized to INTERVENTION MESSAGE #2 and will receive text message reminder (variation #2) about getting their flu shot at their upcoming visit.
  Interventions: Behavioral: Text message reminder
- Cohort 2a (No Intervention): Patients within Cohort 2 do not have an upcoming well visit between September-December 2024, but completed their well visit between January 2023 through August 2024. Patients within Cohort 2a are those randomized to CONTROL and will not receive a text message reminder about getting their flu shot.
- Cohort 2b (Experimental): Patients within Cohort 2 do not have an upcoming well visit between September-December 2024, but completed their well visit between January 2023 through August 2024. Patients within Cohort 2b are those randomized to INTERVENTION MESSAGE #1 and will receive text message reminder (variation #3) about getting their flu shot this upcoming flu season.
  Interventions: Behavioral: Text message reminder
- Cohort 2c (Experimental): Patients within Cohort 2 do not have an upcoming well visit between September-December 2024, but completed their well visit between January 2023 through August 2024. Patients within Cohort 2b are those randomized to INTERVENTION MESSAGE #2 and will receive text message reminder (variation #4) about getting their flu shot this upcoming flu season.
  Interventions: Behavioral: Text message reminder

INTERVENTIONS:
Behavioral: Text message reminder — One-time text message reminder with information about getting flu vaccine at CHOP
  Arms: Cohort 1b; Cohort 1c; Cohort 2b; Cohort 2c

SUMMARY:
Through a large, population-level quality improvement effort within the Children's Hospital of Philadelphia Care Network, we will evaluate text message reminders on flu vaccination rates for both patients with and without a scheduled well child care visit during flu season.

DETAILED DESCRIPTION:
This is a randomized control trial with two patient cohorts: patients with and without a scheduled well child care visit during the upcoming 2024 flu season. Patients with a scheduled well child visit will be randomized into one of three groups (control, intervention message #1, or intervention message #2). Patients within the intervention groups will receive a one-time text message reminder to get their flu shot for their child at their child's upcoming well visit. Intervention groups will be texted at the same time, the same month as their child's well visit. The text message language will differ between groups. Patients without a scheduled upcoming well child visit during the 2024 flu season will also be randomized into one of three groups (control, intervention message #1, or intervention message #2). Intervention groups will be texted at the same time, at the start of flu season. The text message language will differ between groups.

Flu vaccine uptake will be measured within each patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* All patients between ages 6 months-18 years old who have an upcoming well visit during the Fall of 2024 (September through December 2024) or had a completed well visit from January 2023 through August 2024
* Patients have a mobile phone number within their medical record
* Patients have opted-in to text communications from CHOP
* English-speaking

Exclusion Criteria:

* Subjects who do not meet the above inclusion criteria will be excluded

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 228361 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The effectiveness of a text message reminder on influenza vaccine uptake | Baseline to approximately 30 days post-text message
  Via prospective chart review, the primary outcome for both Cohort 1 and Cohort 2 will be to assess the number of patients who received an influenza vaccination 30 days post-text message reminder (baseline). Data from chart review will determine vaccination status (patient received influenza vaccination or not).

SECONDARY OUTCOMES:
The effectiveness of text message language within Cohort 1 | Baseline to approximately 30 days post-text message
  Via prospective chart review, we will compare the number of patients within the Cohort 1 intervention groups who received influenza vaccination to understand which text message variation was more effective. Data from chart review will determine vaccination status (patient received influenza vaccination or not).
The effectiveness of text message language within Cohort 2 | Baseline to approximately 30 days post-text message
  Via prospective chart review, we will compare the number of patients within the Cohort 2 intervention groups who received influenza vaccination to understand which text message variation was more effective. Data from chart review will determine vaccination status (patient received influenza vaccination or not).

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. Jenssen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No